CLINICAL TRIAL: NCT04986462
Title: Arthroscopic Treatment of Bursal-side Partial-thickness Rotator Cuff Tears
Brief Title: Arthroscopic Treatment of Bursal-side Rotator Cuff Tears in Shoulder Joint
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014100
Record Dates: First submitted 2021-06-27; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with bursal-side partial-thickness rotator cuff tears: Patients with bursal-side partial-thickness rotator cuff tears who underwent arthroscopic surgery and was followed up at Peking University Third Hospital.
  Interventions: Procedure: shoulder arthroscopy

INTERVENTIONS:
Procedure: shoulder arthroscopy — Patients underwent ubacromial bursectomy and acromioplasty , cuff debridement and cuff repair, side to side suture of rotator cuff combined with suture anchor.

SUMMARY:
A retrospective analysis was performed on patients with bursal-side partial-thickness rotator cuff tears who underwent arthroscopic surgery from January 2009 to December 2011. To investigate the diagnosis and arthroscopic treatment of partial rotator cuff bursa lateral tear, and to evaluate the postoperative functional outcome and tendon healing.

DETAILED DESCRIPTION:
To study the surgical method and clinical effect of arthroscopic treatment for partial tear of rotator cuff bursa. A retrospective analysis was performed on patients bursal-side partial-thickness rotator cuff tears who underwent arthroscopic surgery from January 2009 to December 2011. Preoperative X-ray and MRI were performed. Rotator cuff repair was performed during the operation. UCLA shoulder scoring scale was used to evaluate the joint at preoperative and final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* From January 2009 to December 2011, patients with bursal-side partial-thickness rotator cuff tears who underwent arthroscopic surgery at Peking University Third Hospital and were followed up.

exclude:

Exclusion Criteria:

* Patients with frozen shoulder and unstable shoulder joints.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bursal-side partial-thickness rotator cuff tears, there has been very little research on bursal-side partial-thickness rotator cuff tears, which has no consensus on diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
UCLA (University of California, Los Angeles) Shoulder Score Scale at 1 year after operation. | 1 year after operation
  Analysis of UCLA (University of California, Los Angeles) Shoulder Score Scale at 1 year after operation. The scale has a minimum score of 2 and a maximum score of 35. The higher the score, the better the prognosis of the patients.
UCLA (University of California, Los Angeles) Shoulder Score Scale at 2 years after operation. | 2 years after operation
  Analysis of UCLA (University of California, Los Angeles) Shoulder Score Scale at 2 years after operation.The scale has a minimum score of 2 and a maximum score of 35. The higher the score, the better the prognosis of the patients.
UCLA (University of California, Los Angeles) Shoulder Score Scale at 5 years after operation. | 5 years after operation
  Analysis of UCLA (University of California, Los Angeles)Shoulder Score Scale at 5 years after operation. The scale has a minimum score of 2 and a maximum score of 35. The higher the score, the better the prognosis of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: jian xiao, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No